CLINICAL TRIAL: NCT03181282
Title: Physical Therapy and Deep Brain Stimulation in Parkinson Disease
Acronym: PTDBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ryan Duncan, Assistant Professor of Physical Therapy, Assistant Professor of Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201609148; K12HD055931 (NIH)
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Balance; Gait; Physical Therapy; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (Experimental): Participants assigned to Physical Therapy (PT) will attend a 1-hour visit with a physical therapist twice weekly for 8 weeks. The PT intervention, which will mirror traditional PT for those with PD, will include exercises designed to improve balance and gait.
  Interventions: Behavioral: Physical Therapy
- Control (No Intervention): Participants in the control group will receive the current standard of care following STN-DBS. As such, STN-DBS settings and anti-PD medications will be optimized according to the determination of their neurologist in the same fashion as they will be in the experimental group. Those in the control group will not receive prescribed exercise from a physical therapist.

INTERVENTIONS:
Behavioral: Physical Therapy — Postural stability exercises will follow a framework targeting quiet stance, anticipatory and reactive postural adjustments, and dynamic postural control. Gait exercises will include treadmill walking and practice with dual-task gait. A home exercise program (HEP), to be completed twice weekly, will be provided on each participant's initial visit with the physical therapist following STN-DBS surgery. The HEP will include the following exercises: trunk rotation, standing hip flexion, standing hip abduction, standing plantarflexion, and standing squat.
  Other Names: Physical Rehabilitation
  Arms: Physical Therapy

SUMMARY:
While deep brain stimulation of the subthalamic nucleus (STN-DBS) is commonly used to reduce tremor, muscle stiffness, and bradykinesia in people with Parkinson disease (PD), preliminary studies suggest balance may worsen and falls may increase after STN-DBS. Walking speed, known to be reduced in PD, typically improves after surgery; however, other important gait qualities may not improve. Given the potential for worsening balance and gait and increasing falls after surgery, it is imperative that researchers explore interventions that complement the positive effects of STN-DBS and delay worsening of balance and gait.

Physical therapy (PT) is reported to be effective in improving balance and walking in people with PD. However, there have been no studies to investigate how individuals with STN-DBS respond to PT. As such, it is unclear if exercise in the post-DBS population is safe, feasible, and effective. The purpose of this study is to examine the safety, feasibility, and efficacy of PT in people with PD with STN-DBS.

The investigators hypothesize that PT will be safe and feasible for people with PD with STN-DBS. Further, the investigators hypothesize that those assigned to PT group will demonstrate improvements in balance and gait while those assigned to the control group will demonstrate no change or a decline in balance and gait.

DETAILED DESCRIPTION:
Deficits in balance and gait may lead to falls, fall-related complications, and physical inactivity in people with PD. These negative effects are thought to lead to a 'malignant' form of PD in which there is reduced quality of life and increased risk for mortality. While people who have had STN-DBS often experience reductions in tremor, rigidity, and bradykinesia, surgical management of PD may not be effective in ameliorating impairments in balance and gait. In fact, investigators have reported that DBS may worsen balance, which may accelerate an individual's decline toward 'malignant' PD. To this end, recent studies indicate physical activity levels did not increase after STN-DBS. This finding should not go unnoticed as physical activity may have a disease modifying effect, slowing the progression of motor disability. As of 2011, approximately 70,000 people with PD have undergone DBS, with the annual number of DBS procedures for PD totaling between 8,000-10,000. In addition, investigators are now studying the effects of STN-DBS in people with early PD. The procedure appears to be safe and effective in this population, which will increase the number of surgical candidates. With the number of people with PD expected to double to more than 8 million by 2030, the number of those receiving DBS is expected to substantially increase.

Given the expected rise in STN-DBS procedures and potential for worsening of postural instability and gait deficits, there is a clear need for interventions that prevent these negative complications of STN-DBS.

Physical therapy, delivered using various treatment approaches (e.g. treadmill training, balance training), is effective in reducing postural instability and improving spatiotemporal gait characteristics among individuals with PD who do not have DBS. To our knowledge, there are no studies to date that assessed the impact of PT for those with PD who have DBS. In fact, the current standard of care following STN-DBS does not include PT. Current care post-DBS includes pharmacologic management and monitoring of DBS settings, which are optimized based on Unified Parkinson's Disease Rating Scale motor subsection (UPDRS III) scores. Despite the introduction of substantial changes to neural activity in areas of the brain governing movement with DBS, formal movement training or assessment of functional mobility and safety are not provided after surgery. As such, patients may not experience significant improvements in postural stability and gait following surgery, and may be at increased risk for falls, fall-related complications, and development of a sedentary lifestyle. Physical therapy is a personalized intervention that can be used to address specific movement impairments that remain even when patients are on optimal regimens of medication and DBS. There is an urgent need to determine if PT is effective in improving postural stability and gait performance over time following STN-DBS. If the intervention is safe and feasible, future studies could evaluate the efficacy of PT for gait and balance deficits in this population before and/or immediately post-surgery, increasing the potential impact of this research.

In this pilot randomized controlled trial, participants will be randomly assigned to either the physical therapy group or control group. Those in the physical therapy group will attend 1-hour sessions of PT twice weekly with a treatment plan designed to improve balance and gait. Those in the control group will not be prescribed an exercise intervention.

Each participant will undergo the same battery of balance and gait tests. Although STN-DBS settings are typically stable at 12 months post-surgery, participants will be allowed to follow up with their neurologists as needed for programming and medication adjustments. All changes in programming settings and medication dosages will be noted. A rater, blinded to group assignment, will collect all outcomes at each time point. Participants will be tested in the following conditions: 1) OFF stimulation and OFF medication and 2) ON stimulation and ON medication. Testing participants OFF stimulation/OFF medication will allow us to determine if the addition of PT after STN-DBS affects balance and gait independent of other treatments. OFF medication is defined as greater than or equal to 12 hours since the last intake of anti-PD medication. For OFF stimulation/OFF medication testing, participants will arrive to the laboratory OFF medication but with stimulators on. The stimulators will be turned OFF upon arrival at the laboratory and testing will commence 45 minutes after the stimulators are turned OFF. Stimulators will be turned back on upon completion of this testing session. The investigators anticipate the total time for this laboratory visit to be 2 hours. Testing ON stimulation/ON medication will provide insight into how participants perform on an everyday basis. ON medication is defined as 1-1.5 hours after medication intake. For ON stimulation/ON medication assessments, participants will arrive to the laboratory 1-1.5 hours after taking their normal anti-PD medication dose with stimulators on and stimulators will remain on throughout the session. Assessments will occur at baseline and at 8 (i.e. post-test) and 12 weeks (i.e. follow up). Assessments will take place on two separate days and the order of testing condition (OFF medication/OFF stimulation vs. ON medication/ON stimulation) will be randomized. The Movement Disorders Society-Unified Parkinson Disease Rating Scale III (MDS-UPDRS III) will be administered in each condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson disease
* Hoehn & Yahr stages II-IV
* At least 1 year post-STN-DBS
* Able to provide informed consent

Exclusion Criteria:

* Diagnosis of atypical parkinsonism
* Hoehn & Yahr stages I or V
* Evidence of dementia (MMSE < 24/30)
* Inability to walk 10 meters with or without assistive device

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Duncan, DPT, Principal Investigator — Washington University in St. Louis School of Medicine - Program in Physical Therapy
Locations (1):
- Washington University in St. Louis School of Medicine - Program in Physical Therapy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duncan RP, Van Dillen LR, Garbutt JM, Earhart GM, Perlmutter JS. Physical therapy and deep brain stimulation in Parkinson's Disease: protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2018 Feb 21;4:54. doi: 10.1186/s40814-018-0243-2. eCollection 2018. PMID 29484198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 participants provided informed consent and were enrolled in the study. 2 participants were unable to complete the baseline assessment and as such were not randomized. 29 participants were randomized to either the intervention or control group.
Pre-assignment Details: The expected enrollment planned for 34 participants due to expected attrition. Due to the lack of attrition, 29 participants were randomized in the study. This corresponds to the power analysis specifying a total sample size of 28 participants.
Period: Overall Study
Arm/Group | Physical Therapy | Control
Started | 15 | 14
Completed | 14 | 14
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Therapy | Control | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (5.8) | 67.8 (7.1) | 65.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 9 | 12 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29
Years Since PD Diagnosis [Mean (Standard Deviation); unit: years] | 12.6 (4.6) | 11.2 (4.9) | 11.9 (4.7)
Months Since STN-DBS [Mean (Standard Deviation); unit: months] | 47.9 (31.2) | 33.9 (27.2) | 41.1 (29.7)
Mini-Mental Status Examination [Median (Full Range); unit: scores on a scale] — The Mini-Mental Status Examination is a global measure of cognitive function. The total possible score ranges from 0 to 30 points. Lower scores indicate worse cognitive function.
  scores on a scale | 28 [25 to 30] | 29 [27 to 30] | 29 [25 to 30]
Movement Disorder Society-Unified Parkinson Disease Rating Scale - Section III (ON) [Mean (Standard Deviation); unit: scores on a scale] — The Movement Disorder Society - Unified Parkinson Disease Rating Scale - Section III is a measure of the severity of motor manifestations of Parkinson disease (PD). The total possible score ranges from 0 to 132 points. Higher scores indicate worsened PD motor severity. The term ON is used to indicate that this measure was obtained when participants were in their clinically optimized state, which means the participants' medication and stimulation were on and working effectively.
  scores on a scale | 36 (13.1) | 30.2 (8.7) | 33.2 (11.4)
Movement Disorder Society-Unified Parkinson Disease Rating Scale - Section III (OFF) [Mean (Standard Deviation); unit: scores on a scale] — The Movement Disorder Society - Unified Parkinson Disease Rating Scale - Section III measures the severity of motor manifestations of Parkinson disease (PD). The total possible score ranges from 0 to 132 points. Higher scores indicate worsened PD motor severity. "OFF" indicates this test was conducted when participants were without medication (>= 12 hours since last dose) and stimulation (stimulators turned off >= 45 minutes before the assessment started). Testing OFF allows assessment of PD manifestations without the influence of medication and stimulation (i.e., true parkinsonian state).
  scores on a scale | 52.1 (11.2) | 46.4 (13.4) | 49.4 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety & Tolerability]
Description: Number of participants with falls, orthopedic injuries, or other adverse events that are related to treatment.
Time Frame: 8 weeks
Population: Because we are interested in potential adverse events related to the the intervention, we assessed only the PT group in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 14 | 0
Participants | 1 |

2. Secondary Outcome: Treatment-Related Adherence [Feasibility]
Description: Feasibility of the treatment as measured by the number of PT sessions attended.
Time Frame: 8 weeks
Population: This variable is analyzed only for the PT group. Because the control group did not attend intervention sessions, this variable is not analyzed for this group.
Measure: Median (Full Range); unit: Number of PT Sessions Attended
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 15 | 0
Number of PT Sessions Attended | 15 [1 to 16] |

3. Secondary Outcome: Balance
Description: Change in Balance Evaluation Systems Test score. The scale is scored from 0-100% with higher scores indicating better balance. Here, the higher the change score, the greater the improvement in balance.
  A change score of 0.04 would correspond to a 4% improvement in the BESTest score. A change score of -0.02 would correspond to a 2% decline in BESTest score.
Time Frame: 8 weeks
Population: For the Off medication / Off stimulation condition, n=13 in the PT group and n=12 in the control group were analyzed. Those not analyzed did not complete this outcome measure at the post-test visit.
Measure: Mean (Standard Deviation); unit: Mean Change in BESTest Percent Score
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 14 | 14
Mean Change in BESTest Percent Score
  On Medication / On Stimulation | 0.04 (0.04) | -0.02 (0.06)
  Off Medication / Off Stimulation: number analyzed (Participants) | 13 | 12
  Off Medication / Off Stimulation | 0.03 (0.05) | -0.04 (0.07)
Statistical Analysis 1: Comparison: Physical Therapy vs Control; This analysis is for the On Medication / On Stimulation condition. Age was controlled for in the analysis given the baseline difference in age between groups; Test type: Superiority; p = 0.0194, Mixed Models Analysis; Mixed model analysis with repeated measures; Slope = 0.0529, 95% CI 2-sided [0.0132 to 0.0925], Standard Error of Mean 0.0194
Statistical Analysis 2: Comparison: Physical Therapy vs Control; This analysis is for the Off Medication / Off Stimulation Condition. Age was controlled for in the analysis given the baseline difference in age between groups; Test type: Superiority; p = 0.004625, Mixed Models Analysis; Mixed models analysis with repeated measures; Slope = 0.0718, 95% CI 2-sided [0.0242 to 0.1194], Standard Error of Mean 0.0231

4. Secondary Outcome: Gait
Description: Change in gait velocity (cm/sec). Higher gait speeds are associated with better mobility. The greater the value for the change in gait speed, the greater the improvement in gait speed. Negative values would indicate a decline in gait speed.
Time Frame: 8 weeks
Population: For the Off medication / Off stimulation analysis, n=14 in the PT group and n=12 in the control group were analyzed. Those not analyzed did not complete this outcome measure at the post-test visit.
Measure: Mean (Standard Deviation); unit: Change in Gait Velocity (Cm/Sec)
Arm/Group | Physical Therapy | Control
Number analyzed (Participants) | 14 | 14
Change in Gait Velocity (Cm/Sec)
  On Medication / On Stimulation | 9.71 (15.02) | -1.07 (10.5)
  Off Medication / Off Stimulation: number analyzed (Participants) | 14 | 12
  Off Medication / Off Stimulation | 7.29 (12.84) | -1.00 (11.05)
Statistical Analysis 1: Comparison: Physical Therapy vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.038389, Mixed Models Analysis; Mixed models analysis with repeated measures; Slope = 10.5248, 95% CI 2-sided [0.6038 to 20.4459], Standard Error of Mean 4.8439
Statistical Analysis 2: Comparison: Physical Therapy vs Control; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.109873, Mixed Models Analysis; Mixed models analysis with repeated measures; Slope = 7.7233, 95% CI 2-sided [-1.8652 to 17.3117], Standard Error of Mean 4.6680

ADVERSE EVENTS:
Time Frame: The time frame of interest for adverse events was 8 weeks (after completion or pre-test and just prior to completion of post-test assessments).
Description: Adverse events were collected weekly via phone interview using a custom questionnaire.
Arm/Group | Physical Therapy | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/14
Other Adverse Events (participants affected / at risk) | 10/15 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Therapy (N=15) | Control (N=14)
Chest Pain (Cardiac disorders) | 1 (1) | 2 (3) — One participant in the PT group had 1 episode of chest pain that occurred outside PT treatment. A cardiac stent was placed. Two participants in the control group reported chest pain. These reports were determined to be not of cardiac origin.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Therapy (N=15) | Control (N=14)
Fall (Nervous system disorders) | 9 (35) | 9 (19) — The falls occurred outside of the PT intervention.
Severe Joint Pain (Musculoskeletal and connective tissue disorders) | 8 (40) | 5 (15) — Reports of severe joint pain were associated with pain that preceded study participation (PT group) or occurred in the control group (unrelated to intervention). Severe joint pain was recorded as one event/week regardless of the number of locations.
Persistent Muscle Soreness (> 2 days) (Musculoskeletal and connective tissue disorders) | 8 (21) | 6 (21) — Persistent muscle soreness was recorded as one event/week regardless of the number of locations.
Dizziness/Lightheaded (Nervous system disorders) | 1 (1) | 4 (11) — Participant reports of feeling dizzy or lightheaded.
Extreme Fatigue (Nervous system disorders) | 0 (0) | 4 (10) — Reports of extreme fatigue.
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Reports of muscle cramping.
Common Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Reports of symptoms related to the common cold (e.g., cough).
Anxiety Attack (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Muscle Pain/Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tooth Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Foot Soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral Elbow Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tricep Nerve Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eye Infection (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a small trial with a small number of participants. The intervention lasted only 8 weeks. Further, there were baseline differences between the groups that should be considered when interpreting the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03181282/Prot_SAP_000.pdf